CLINICAL TRIAL: NCT02083536
Title: A Phase I Study Using Low-Dose Fractionated Whole Abdominal Radiation Therapy (LDFWART) As A Docetaxel Chemo-Potentiator for Patients With Platinum-Resistant Recurrent Ovarian Carcinoma
Brief Title: LDFWART With Docetaxel in Patients With Platinum-Resistant Recurrent Ovarian Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study voluntarily stopped by Principal Investigator due to lack of accrual.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Aaron Wolfson, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110671
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Recurrent Ovarian Cancer; Recurrent Ovarian Carcinoma
Keywords: Low Dose Fractionated Whole Abdominal Radiation Therapy; LDFWART; Docetaxel; Ovarian Cancer; Ovarian Carcinoma; Platinum-Resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDFWART + Docetaxel (Experimental): This study has 6 treatment cycles given at 3 weeks intervals ± 3 days. A cycle is defined as 1 treatment of morning Docetaxel and afternoon Low Dose Fractionated Whole Abdominal Radiation Therapy (LDFWART). The first day of the first treatment is designated "study day 1".
  Interventions: Radiation: Low Dose Fractionated Whole Abdominal Radiation Therapy; Drug: Docetaxel

INTERVENTIONS:
Radiation: Low Dose Fractionated Whole Abdominal Radiation Therapy — A single fraction of LDFWART will be given 6-8 hours after the start of morning administration of Docetaxel for 6 cycles (the time of the start Docetaxel will be counted as the frame of reference for when the LDFWART can be given).
  Other Names: LDFWART
Drug: Docetaxel — Chemotherapy will consist of 6 cycles of Docetaxel. Each cycle will follow standard of care and will be scheduled every 3 weeks ± 3 days. Chemotherapy should be administered in the morning to allow 6-8 hours before Radiation Therapy. On Day 1 of each cycle, chemotherapy will consist of Docetaxel 60 mg/m² infused intravenously over 30-60 minutes (with premedication of dexamethasone 10 mg given IV 30-60 minutes prior to docetaxel administration).
  Other Names: Taxotere

SUMMARY:
The ultimate clinical aim of this proposed phase I trial is to evaluate the toxicity and determine the recommended phase II dose of combining the effect of LDFWART following administration of docetaxel for 6 cycles in patients with recurrent platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have platinum-resistant disease relapsing within 6 months or less from the date of their last cycle of initial adjuvant chemotherapy recurrent adenocarcinoma from a primary ovarian, tubal, or peritoneal cancer following first-line chemotherapy for metastatic disease. There is no limit on prior number of chemotherapy regimens. Patients who have received prior systemic docetaxel and platinum-based chemotherapy are eligible
* 1.1 Patients must have ≥ 1cm measurable disease on imaging studies independent of patients having an optional surgical salvage procedure.
* 2. Patients must have a life expectancy of at least 6 months.
* 3. Patients must have Karnofsky performance status of ≥ 60 or Gynecology Oncology (GOG) performance status of ≤ 2 (see www.GOG.org website).
* 4. Age 18 - 80 years old
* 5. Patients must have an adequate bone marrow, renal, and hepatic function:

  * 5.1 WBC: ≥ 3,000 /mcl
  * 5.2 ANC: ≥ 1,500 /mcl
  * 5.3 Platelets: ≥ 100,000 /mcl
  * 5.4 Creatinine: < 2.0 mg/dcl
  * 5.5 Bilirubin: < 1.5x institutional normal value
  * 5.6 LDH, GGT, SGPT (ALT), SGOT (AST), and ALK Phos:< 3x institutional normal value.
* 6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* 1. Patients who have received prior radiotherapy to the chest, whole abdomen, or lower extremities above the knees.
* 2. Patients who have received prior radiation therapy to the head, neck, or lower extremities below the knees if greater than 3 years prior to study entry.
* 3. Evidence of extra-abdominal extension of disease (such as groin nodes, lung, supraclavicular nodes, and pleural fluid).
* 4. Patients may not be receiving any other investigational agents within 4 weeks preceding the start of study treatment) or chemotherapy for at least 3 weeks preceding the start of study treatment.
* 5. Patients who have been diagnosed with another prior malignant tumor within 3 years of study entry, excluding non-melanoma skin cancer and carcinoma in situ of the cervix.
* 6. Patients with prior history of a severe hypersensitivity reaction to paclitaxel (polysorbate 80-Cremophor).
* 7. Patients with current history of uncontrolled hypertension, angina pectoris, heart failure, cardiac dysrhythmias, pericardial disease, cardiomyopathy, or active infection.
* 8. Presence of any medical condition that in the opinion of the investigator deems the patient unable to participate.
* 9. Females of child-bearing potential. It is expected that ovarian cancer patients would have had a hysterectomy and/or oophorectomy as part of the original standard of care.
* 10. Patients that are < 18 yrs. of age or > 80 yrs. of age.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Adverse Events as a Measure of Safety and Tolerability | 3 years
  Number of subjects experiencing adverse events after receiving protocol therapy.
Recommended Phase II Dose of LDFWART | 3 years
  The recommended phase II dose of low-dose whole abdominal radiation therapy (LDFWART) when used in conjunction with 6 cycles of docetaxel chemotherapy.

SECONDARY OUTCOMES:
Number of Subjects Experiencing Complete or Partial Response to Protocol Therapy | Up to 5 years
  Number of subjects experiencing complete response (CR) or partial response (PR) according to RECIST Criteria Version 1.1
The rate of Overall Survival in subjects receiving protocol therapy | Up to 5 years
  Observed length of life from start of treatment to cause of death
The rate of Progression-Free Survival in subjects receiving protocol therapy. | Up to 5 years
  Length of time from start of treatment to the time of documented disease progression in study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H Wolfson, MD, Principal Investigator — University of Miami